CLINICAL TRIAL: NCT04811300
Title: A Single-Center, Prospective Clinical Study to Demonstrate That in 4 Different Lighting Conditions mCVI® Accurately Captures Pulse Rate and Respiratory Rate in 10 Healthy Volunteers in Comparison to a Commercially-Available Masimo Pulse Oximeter Device
Brief Title: mCVI® Lighting Conditions Clinical Study
Status: Completed | Type: Observational
Sponsor: Intelomed, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: mCVI003
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Algorithm Verification

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: There is no intervention — There is no intervention

SUMMARY:
This single center prospective clinical study is to verify the algorithm of mCVI® in 4 different lighting conditions to accurately capture pulse rate and respiratory rate in 10 healthy subjects in comparison to commercially-available Masimo pulse oximeter devices. This is a non significant risk device.

DETAILED DESCRIPTION:
In this prospective clinical study the mCVI® device is a mobile application used to simply verify the algorithm when the mobile video reads a patients pulse rate and respiratory rate while spontaneously breathing. There is no facial recognition technology. There is no immediate feedback given to the research team to act upon or provide for further clinical care decisions. In real time, the mCVI® device will be compared to two commercially-available Masimo pulse oximeter devices in a single visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between the ages of 21 - 70
* Informed consent obtained and signed

Exclusion Criteria:

* Self-reported medical conditions that could compromise a participant's ability to provide for all breathing samples, pedal the Cubii Pro elliptical, or follow instructions
* Self-reported medical history of respiratory or cardiovascular disease
* Excessive facial hair, facial deformities, or obstructions (like glasses or face masks/shields) that could compromise the recording of pulse rate and respiratory rate of the mCVI®
* Any face lotions or make up foundations that could compromise the recording of pulse rate and respiration rate of the mCVI®
* Missing digits or fingers on one or more hand that would prevent proper recording of Masimo pulse oximeter devices
* Participants wearing nail polish, acrylic nails, or rings on the ring finger of either hand that would prevent the proper use of Masimo pulse oximeter device
* Inability to provide informed consent

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2021-04-11 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Pulse Rate Verification in Different Lighting Conditions | 2 months
  To demonstrate that in 4 different lighting environments common to home and office/clinical conditions, mCVI® accurately captures pulse rate in comparison to Masimo pulse oximeter devices.
Respiration Rate Verification in Different Lighting Conditions | 2 months
  To demonstrate that in 4 different lighting environments common to home and office/clinical conditions, mCVI® accurately captures respiratory rate in comparison to Masimo pulse oximeter devices.

SECONDARY OUTCOMES:
Skin Tone Pulse Rate Verification in Different Lighting Conditions | 2 months
  To demonstrate that in 4 different lighting environments common to home and office/clinical conditions, mCVI® accurately captures pulse rate in healthy volunteers with a variety of skin tones using the Fitzpatrick Skin Type Scale.
Skin Tone Respiratory Rate Verification in Different Lighting Conditions | 2 months
  To demonstrate that in 4 different lighting environments common to home and office/clinical conditions, mCVI® accurately captures respiration rates in healthy volunteers with a variety of skin tones using the Fitzpatrick Skin Type Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Scitech Campus Corporation, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No